CLINICAL TRIAL: NCT06452134
Title: Evaluation the Effect of Coenzyme Q10 on Tissue Healing Process in Patients Undergoing Wisdom Tooth Extraction in the City of Sanandaj-Iran in 1402: a Double-blinded Clinical Trial Study
Brief Title: Evaluation the Effect of Coenzyme Q10 on Tissue Healing Process in Patients Undergoing Wisdom Tooth Extraction
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Zahra Nejati (Other)
Collaborators: Kurdistan University of Medical Sciences (Other); Hady Mohammadi, Director of oral and maxillofacial surgery department, school of dentistry, Kurdistan university of medical sciences (Unknown); Yousef Moradi, Assistant professor, Department of epidemiology and biostatistics, Kurdistan university of medical sciences (Unknown); Babak Ghadirzadeh, medical student, Kurdistan university of medical sciences (Unknown)
Responsible Party: Sponsor-Investigator, Zahra Nejati, Zahra Nejati, Dental student, Department of oral and maxillofacial medicine, School of Dentistry, Kurdistan University of Medical Sciences, Sanandaj, Iran., Kurdistan University of Medical Sciences
Organization: Kurdistan University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IR.MUK.REC.1403.030
Record Dates: First submitted 2024-05-30; First posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Molar, Third; Temporomandibular Joint Disorders; Dry Socket; Coenzyme Q10
Keywords: coenzyme Q10; Dry Socket; Temporomandibular Joint Disorders; Molar, Third; SF-36 health survey; Tissue healing; Tooth Extraction; GHQ-12
MeSH Terms: conditions — Temporomandibular Joint Disorders; Dry Socket | interventions — coenzyme Q10; Tablets; Ubiquinone

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): This arm of the study includes 35 of participants who will be given Coenzyme Q10 100 MG Oral Tablet for 30 days.
  Interventions: Drug: Coenzyme Q10 100 MG Oral Tablet
- Control group (Placebo Comparator): This arm of the study includes 35 of participants who will be given Placebo ( a look-alike substance ) with same tablet form given daily for a period of 30 days after surgery.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Coenzyme Q10 100 MG Oral Tablet — Coenzyme Q10 oral Tablet with dosage of 100mg daily given for a period of 30 days after surgery.
  Other Names: Coenzyme Q; CoQ; CoQ10; Ubiquinone; Ubiquinone-Q10; Ubidecarenone; Vitamin Q10
  Arms: Intervention group
Drug: Placebo — Exactly same looking agent in the form of a tablet with same size and color to CoezymeQ10 with no active property given for a period of 30 days after surgery.
  Arms: Control group

SUMMARY:
The goal of this clinical trial is to asses the effect of Coenzyme Q10 administration in patients from any gender group who are older than 18 years old undergoing wisdom tooth extraction. The main questions it aims to answer are:

does Coenzyme Q10 help with better tissue healing? does Coenzyme Q10 administration lower the prevalence of Dry socket after surgery? does Coenzyme Q10 prevent TMD (Temporomandibular disorders) while recovering from surgery? how does Coenzyme Q10 administration effect the answers to SF-36 health survey in patients? Researchers will compare Coenzyme Q10 to a placebo (a look-alike substance that contains no drug) to see if it has any effect on mentioned parameters.

Participants will:

* take coenzyme Q10 (100mg) daily for 30 days after surgery.
* will be examined and evaluated 1, 7, 14 and 30 days after completion of surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years old that require mandibular or maxillary molar, third tooth extraction as Oral and Maxillofacial surgeon's clinical diagnosis.

Exclusion Criteria:

* The patient's departure from Sanandaj
* The patient's disagreement with the study protocol
* The Patient's demise
* The patient's hospitalization for unrelated illnesses
* The patient's discontent with the care they received
* The patient's failure to show up for follow-up appointments
* The patient's sensitivity to Coenzyme Q10

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Rate of Tissue healing | 1, 7, 14 and 30 days after surgery
  Regeneration-the replacement of damaged tissues with cells of the same type-and fibrosis-the replacement of damaged tissues with connective tissue-are the two primary processes involved in wound healing. To help in tissue healing, some cells, such as fibroblasts and vascular endothelial cells, have the ability to proliferate quickly in response to an external stimulation. Wound closure also requires non-proliferating cells, such as peripheral nervous system cells and odontoblasts. The bone that grows in to fill the space left by a tooth extraction should be similar to the surrounding healthy tissues. A lack of tissue healing is indicated by symptoms such as edema, fever, bleeding, discomfort, necrosis, exudate, flap instability, foul taste, and fistula. If trismus results from a muscle injury following an IAN Block injection, it should go away as the tissue heals.

SECONDARY OUTCOMES:
Incidence of Temporomandibular disorders | 1, 7, 14 and 30 days after surgery
  Temporomandibular disorders is a collective term for a set of disorders characterized by pain and dysfunction in the muscles and jaw joint. A specialist dentist will measure a patient's temporomandibular disorder (TMD) clinically by looking for signs of trismus, abnormal movement of the lower jaw during opening and closing or chewing, jaw dysfunction, reduced range of motion, ear pain, temporal pain, headache, bruxism, sensitivity of the muscles in the neck and shoulders, and malocclusion (such as acquired edentulism, facial asymmetry, etc.). The diagnosis of TMD is finalized if the symptoms are positive.
Occurrence of Dry socket | 1, 7, 14 and 30 days after surgery
  This is a non-scientific phrase for a cavity where all or part of the bone is exposed since there isn't any bone in the days following extraction. This can happen inside the cavity or outside the occlusal environment of the cavity. Severe recurrent pain results from the patient's inability to stop the mechanical stimulation of food particles or tongue on the exposed bone, which is extremely painful to touch. A specialized physician measures it by doing a clinical examination as well as by observing the whiteness of the bone-which is empty and uncomfortable to the touch-in the extracted tooth's socket.
Answers to The Short Form Health Survey-36 | 1, 7, 14 and 30 days after surgery
  This tool has shown to be useful in a variety of contexts, including clinical practice, the assessment of health policies, and general security investigations. The 36-item form was created in the United States in 1992 by Ware and associates, and studies on a range of patient populations have assessed its validity and reliability. This questionnaire's topics are not restricted to any one age range, illness, or condition. By adding the results of the eight health-forming categories, the questionnaire's design aims to assess the state of health from both a physical and mental standpoint. This survey, which consists of 63 items, rates eight distinct health domains using a scoring system derived from the table found in the reference. To score the SF-36, scales are standardized with a scoring algorithm or by the SF-36v2 scoring software to obtain a score ranging from 0 to 100. Higher scores indicate better health status.
Answers to The General Health Questionnaire-12 | 1, 7, 14 and 30 days after surgery
  Developed in the 1970s, the General Health Questionnaire (GHQ) is regarded as a valid and dependable instrument for evaluating mental health. The most popular of the various iterations of this survey is the GHQ-12 version. It is a 12-item mental health assessment that is assessed using the table given in the reference.The scores typically used are the binary scale (0-0-1-1) and the 4-point Likert-type scale (0-1-2-3). Responses to all items are summed up to a total score ranging from 0 to 12 (binary scale) or 0 to 36 (Likert scale), with higher scores indicating more severe impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Zahra Nejati, Study Director — Zahra Nejati, Department of oral and maxillofacial medicine, School of Dentistry, Kurdistan University of Medical Sciences, Sanandaj, Iran.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rafetto LK. Managing Impacted Third Molars. Oral Maxillofac Surg Clin North Am. 2015 Aug;27(3):363-71. doi: 10.1016/j.coms.2015.04.004. Epub 2015 Jun 9. PMID 26070801
- [Result] Glickman A, Karlis V. Pediatric Benign Soft Tissue Oral and Maxillofacial Pathology. Oral Maxillofac Surg Clin North Am. 2016 Feb;28(1):1-10. doi: 10.1016/j.coms.2015.07.005. PMID 26614696
- [Result] Kaner KH. Referral and Management Considerations for a Biopsy: Why Choose the Oral and Maxillofacial Surgeon. Dent Clin North Am. 2020 Jan;64(1):241-247. doi: 10.1016/j.cden.2019.08.013. Epub 2019 Oct 21. PMID 31735229
- [Result] Kiencalo A, Jamka-Kasprzyk M, Panas M, Wyszynska-Pawelec G. Analysis of complications after the removal of 339 third molars. Dent Med Probl. 2021 Jan-Mar;58(1):75-80. doi: 10.17219/dmp/127028. PMID 33789003
- [Result] Hallab L, Azzouzi A, Chami B. Quality of life after extraction of mandibular wisdom teeth: A systematic review. Ann Med Surg (Lond). 2022 Aug 21;81:104387. doi: 10.1016/j.amsu.2022.104387. eCollection 2022 Sep. PMID 36147052
- [Result] Hao M, Duan M, Yang Z, Zhou H, Li S, Xiang J, Wu H, Liu H, Chang L, Wang D, Liu W. Engineered stem cell exosomes for oral and maxillofacial wound healing. Front Bioeng Biotechnol. 2022 Oct 24;10:1038261. doi: 10.3389/fbioe.2022.1038261. eCollection 2022. PMID 36353739
- [Result] Cluis CP, Burja AM, Martin VJ. Current prospects for the production of coenzyme Q10 in microbes. Trends Biotechnol. 2007 Nov;25(11):514-21. doi: 10.1016/j.tibtech.2007.08.008. PMID 17935805
- [Result] Moon HJ, Ko WK, Han SW, Kim DS, Hwang YS, Park HK, Kwon IK. Antioxidants, like coenzyme Q10, selenite, and curcumin, inhibited osteoclast differentiation by suppressing reactive oxygen species generation. Biochem Biophys Res Commun. 2012 Feb 10;418(2):247-53. doi: 10.1016/j.bbrc.2012.01.005. Epub 2012 Jan 9. PMID 22252298
- [Result] Sifuentes-Franco S, Sanchez-Macias DC, Carrillo-Ibarra S, Rivera-Valdes JJ, Zuniga LY, Sanchez-Lopez VA. Antioxidant and Anti-Inflammatory Effects of Coenzyme Q10 Supplementation on Infectious Diseases. Healthcare (Basel). 2022 Mar 7;10(3):487. doi: 10.3390/healthcare10030487. PMID 35326965
- [Result] Li X, Zhan J, Hou Y, Hou Y, Chen S, Luo D, Luan J, Wang L, Lin D. Coenzyme Q10 Regulation of Apoptosis and Oxidative Stress in H2O2 Induced BMSC Death by Modulating the Nrf-2/NQO-1 Signaling Pathway and Its Application in a Model of Spinal Cord Injury. Oxid Med Cell Longev. 2019 Dec 12;2019:6493081. doi: 10.1155/2019/6493081. eCollection 2019. PMID 31915512
- [Result] Hargreaves I, Heaton RA, Mantle D. Disorders of Human Coenzyme Q10 Metabolism: An Overview. Int J Mol Sci. 2020 Sep 13;21(18):6695. doi: 10.3390/ijms21186695. PMID 32933108
- [Result] Moon HJ, Ko WK, Jung MS, Kim JH, Lee WJ, Park KS, Heo JK, Bang JB, Kwon IK. Coenzyme q10 regulates osteoclast and osteoblast differentiation. J Food Sci. 2013 May;78(5):H785-891. doi: 10.1111/1750-3841.12116. Epub 2013 Apr 12. PMID 23582186
- [Result] Kaushik AS, Strath LJ, Sorge RE. Dietary Interventions for Treatment of Chronic Pain: Oxidative Stress and Inflammation. Pain Ther. 2020 Dec;9(2):487-498. doi: 10.1007/s40122-020-00200-5. Epub 2020 Oct 21. PMID 33085012
- [Result] Bonakdar RA, Guarneri E. Coenzyme Q10. Am Fam Physician. 2005 Sep 15;72(6):1065-70. PMID 16190504
- [Result] Choi BS, Song HS, Kim HR, Park TW, Kim TD, Cho BJ, Kim CJ, Sim SS. Effect of coenzyme Q10 on cutaneous healing in skin-incised mice. Arch Pharm Res. 2009 Jun;32(6):907-13. doi: 10.1007/s12272-009-1613-3. Epub 2009 Jun 26. PMID 19557369
- [Result] Mencucci R, Favuzza E, Boccalini C, Lapucci A, Felici R, Resta F, Chiarugi A, Cavone L. CoQ10-containing eye drops prevent UVB-induced cornea cell damage and increase cornea wound healing by preserving mitochondrial function. Invest Ophthalmol Vis Sci. 2014 Oct 9;55(11):7266-71. doi: 10.1167/iovs.14-15306. PMID 25301877
- [Result] Gulsen I, Ak H, Colcimen N, Alp HH, Akyol ME, Demir I, Atalay T, Balahroglu R, Ragbetli MC. Neuroprotective Effects of Thymoquinone on the Hippocampus in a Rat Model of Traumatic Brain Injury. World Neurosurg. 2016 Feb;86:243-9. doi: 10.1016/j.wneu.2015.09.052. Epub 2015 Sep 30. PMID 26428323
- [Result] Manzar H, Abdulhussein D, Yap TE, Cordeiro MF. Cellular Consequences of Coenzyme Q10 Deficiency in Neurodegeneration of the Retina and Brain. Int J Mol Sci. 2020 Dec 6;21(23):9299. doi: 10.3390/ijms21239299. PMID 33291255
- [Result] Al Saadi T, Assaf Y, Farwati M, Turkmani K, Al-Mouakeh A, Shebli B, Khoja M, Essali A, Madmani ME. Coenzyme Q10 for heart failure. Cochrane Database Syst Rev. 2021 Feb 3;(2)(2):CD008684. doi: 10.1002/14651858.CD008684.pub3. PMID 35608922
- [Result] Abdelkader HA, Rashed LA, Assaad E, Saleh MA. Serum and tissue levels of coenzyme Q10 in pemphigus vulgaris. J Cosmet Dermatol. 2022 Jul;21(7):3002-3006. doi: 10.1111/jocd.14511. Epub 2021 Oct 3. PMID 34601804
- [Result] Ghasemi S, Torab Z, Shirmohammadi A, Babaloo A, Johari R, Farhadi F, Mobasseri M, Mohammadi H. Evaluation of the effect of coenzyme Q10 supplementation along with scaling and root planing (SRP) on periodontal and gingival indices in controlled diabetic patients. J Adv Periodontol Implant Dent. 2022 Mar 13;14(1):32-37. doi: 10.34172/japid.2022.003. eCollection 2022. PMID 35919443
- [Result] Ko KI, Sculean A, Graves DT. Diabetic wound healing in soft and hard oral tissues. Transl Res. 2021 Oct;236:72-86. doi: 10.1016/j.trsl.2021.05.001. Epub 2021 May 13. PMID 33992825
- [Result] Marini L, Rojas MA, Sahrmann P, Aghazada R, Pilloni A. Early Wound Healing Score: a system to evaluate the early healing of periodontal soft tissue wounds. J Periodontal Implant Sci. 2018 Oct 24;48(5):274-283. doi: 10.5051/jpis.2018.48.5.274. eCollection 2018 Oct. PMID 30405935
- [Result] List T, Jensen RH. Temporomandibular disorders: Old ideas and new concepts. Cephalalgia. 2017 Jun;37(7):692-704. doi: 10.1177/0333102416686302. Epub 2017 Jan 9. PMID 28068790
- [Result] Bowe DC, Rogers S, Stassen LF. The management of dry socket/alveolar osteitis. J Ir Dent Assoc. 2011 Dec-2012 Jan;57(6):305-10. PMID 22338284
- [Result] Reale C, Invernizzi F, Panteghini C, Garavaglia B. Genetics, sex, and gender. J Neurosci Res. 2023 May;101(5):553-562. doi: 10.1002/jnr.24945. Epub 2021 Sep 9. PMID 34498752
- [Result] Newland JA. How do you define age? Nurse Pract. 2014 Jul 13;39(7):6. doi: 10.1097/01.NPR.0000450740.92453.2b. No abstract available. PMID 24878832
- [Result] Bailey E, Kashbour W, Shah N, Worthington HV, Renton TF, Coulthard P. Surgical techniques for the removal of mandibular wisdom teeth. Cochrane Database Syst Rev. 2020 Jul 26;7(7):CD004345. doi: 10.1002/14651858.CD004345.pub3. PMID 32712962
- [Result] Miloro M, DaBell J. Radiographic proximity of the mandibular third molar to the inferior alveolar canal. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2005 Nov;100(5):545-9. doi: 10.1016/j.tripleo.2005.03.009. PMID 16243238
- [Result] Fry RR, Patidar DC, Goyal S, Malhotra A. Proximity of maxillary posterior teeth roots to maxillary sinus and adjacent structures using Denta scan(R). Indian J Dent. 2016 Sep;7(3):126-130. doi: 10.4103/0975-962X.189339. PMID 27795646
- [Result] Dodson TB, Susarla SM. Impacted wisdom teeth. BMJ Clin Evid. 2014 Aug 29;2014:1302. PMID 25170946
- [Result] Unwerawattana W. Common symptoms and type of impacted molar tooth in King Chulalongkorn Memorial Hospital. J Med Assoc Thai. 2006 Sep;89 Suppl 3:S134-9. PMID 17718279
- [Result] Doty RL. Systemic diseases and disorders. Handb Clin Neurol. 2019;164:361-387. doi: 10.1016/B978-0-444-63855-7.00021-6. PMID 31604558
- [Result] Dean E. Anxiety. Nurs Stand. 2016 Jul 13;30(46):15. doi: 10.7748/ns.30.46.15.s17. PMID 27406490
- [Result] Al-Qudah AA, Bani Younis HAB, Awawdeh LA, Daud A. Root and canal morphology of third molar teeth. Sci Rep. 2023 Apr 27;13(1):6901. doi: 10.1038/s41598-023-34134-7. PMID 37106025
- [Result] Mehrotra N, Singh S. Periodontitis. 2023 May 1. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK541126/ PMID 31082170
- [Result] Dolens Eda S, Nakai FV, Santos Parizi JL, Alborghetti Nai G. Cytopathology: a useful technique for diagnosing oral lesions?: a systematic literature review. Diagn Cytopathol. 2013 Jun;41(6):505-14. doi: 10.1002/dc.22875. Epub 2012 May 30. PMID 22645047
- [Result] Yaseen SM, Naik S, Uloopi KS. Ectopic eruption - A review and case report. Contemp Clin Dent. 2011 Jan;2(1):3-7. doi: 10.4103/0976-237X.79289. PMID 22114445
- [Result] Esian D, Bica CI, Stoica OE, Dako T, Vlasa A, Bud ES, Salcudean D, Beresescu L. Prevalence and Manifestations of Dental Ankylosis in Primary Molars Using Panoramic X-rays: A Cross-Sectional Study. Children (Basel). 2022 Aug 8;9(8):1188. doi: 10.3390/children9081188. PMID 36010078
- [Result] van Lummel RC, Walgaard S, Pijnappels M, Elders PJ, Garcia-Aymerich J, van Dieen JH, Beek PJ. Physical Performance and Physical Activity in Older Adults: Associated but Separate Domains of Physical Function in Old Age. PLoS One. 2015 Dec 2;10(12):e0144048. doi: 10.1371/journal.pone.0144048. eCollection 2015. PMID 26630268
- [Result] Montazeri A, Goshtasebi A, Vahdaninia M, Gandek B. The Short Form Health Survey (SF-36): translation and validation study of the Iranian version. Qual Life Res. 2005 Apr;14(3):875-82. doi: 10.1007/s11136-004-1014-5. PMID 16022079
- [Result] Masciocchi E, Maltais M, El Haddad K, Virecoulon Giudici K, Rolland Y, Vellas B, de Souto Barreto P. Defining Vitality Using Physical and Mental Well-Being Measures in Nursing Homes: A Prospective Study. J Nutr Health Aging. 2020;24(1):37-42. doi: 10.1007/s12603-019-1285-8. PMID 31886806
- [Result] Cohen M, Quintner J, van Rysewyk S. Reconsidering the International Association for the Study of Pain definition of pain. Pain Rep. 2018 Mar 5;3(2):e634. doi: 10.1097/PR9.0000000000000634. eCollection 2018 Mar. PMID 29756084
- [Result] Brussow H. What is health? Microb Biotechnol. 2013 Jul;6(4):341-8. doi: 10.1111/1751-7915.12063. Epub 2013 May 6. PMID 23647782
- [Result] Riley RD, Ensor J, Snell KIE, Harrell FE Jr, Martin GP, Reitsma JB, Moons KGM, Collins G, van Smeden M. Calculating the sample size required for developing a clinical prediction model. BMJ. 2020 Mar 18;368:m441. doi: 10.1136/bmj.m441. No abstract available. PMID 32188600
- [Result] Zhong B. How to calculate sample size in randomized controlled trial? J Thorac Dis. 2009 Dec;1(1):51-4. PMID 22263004
- [Result] Althunian TA, de Boer A, Groenwold RHH, Klungel OH. Defining the noninferiority margin and analysing noninferiority: An overview. Br J Clin Pharmacol. 2017 Aug;83(8):1636-1642. doi: 10.1111/bcp.13280. Epub 2017 Apr 6. PMID 28252213
- [Result] Sakpal TV. Sample size estimation in clinical trial. Perspect Clin Res. 2010 Apr;1(2):67-9. PMID 21829786
- [Result] Lachin JM, Matts JP, Wei LJ. Randomization in clinical trials: conclusions and recommendations. Control Clin Trials. 1988 Dec;9(4):365-74. doi: 10.1016/0197-2456(88)90049-9. PMID 3203526
- [Result] Berger VW, Bour LJ, Carter K, Chipman JJ, Everett CC, Heussen N, Hewitt C, Hilgers RD, Luo YA, Renteria J, Ryeznik Y, Sverdlov O, Uschner D; Randomization Innovative Design Scientific Working Group. A roadmap to using randomization in clinical trials. BMC Med Res Methodol. 2021 Aug 16;21(1):168. doi: 10.1186/s12874-021-01303-z. PMID 34399696
- [Result] Pippi R. Post-Surgical Clinical Monitoring of Soft Tissue Wound Healing in Periodontal and Implant Surgery. Int J Med Sci. 2017 Jul 18;14(8):721-728. doi: 10.7150/ijms.19727. eCollection 2017. PMID 28824306
- [Result] Zwahlen RA, Cheung LK, Zheng LW, Chow RL, Li T, Schuknecht B, Gratz KW, Weber FE. Comparison of two resorbable membrane systems in bone regeneration after removal of wisdom teeth: a randomized-controlled clinical pilot study. Clin Oral Implants Res. 2009 Oct;20(10):1084-91. doi: 10.1111/j.1600-0501.2009.01751.x. PMID 19751357
- [Result] Covani U, Barone A, Cornelini R, Crespi R. Soft tissue healing around implants placed immediately after tooth extraction without incision: a clinical report. Int J Oral Maxillofac Implants. 2004 Jul-Aug;19(4):549-53. PMID 15346752
- [Result] Gauer RL, Semidey MJ. Diagnosis and treatment of temporomandibular disorders. Am Fam Physician. 2015 Mar 15;91(6):378-86. PMID 25822556
- [Result] Mamoun J. Dry Socket Etiology, Diagnosis, and Clinical Treatment Techniques. J Korean Assoc Oral Maxillofac Surg. 2018 Apr;44(2):52-58. doi: 10.5125/jkaoms.2018.44.2.52. Epub 2018 Apr 25. PMID 29732309
- [Result] Keselman HJ, Algina J, Kowalchuk RK. The analysis of repeated measures designs: a review. Br J Math Stat Psychol. 2001 May;54(Pt 1):1-20. doi: 10.1348/000711001159357. PMID 11393894
- [Derived] Nejati Z, Ghadirzadeh B, Mohammadi H, Afraie M, Moradi Y. Effect of coenzyme Q10 on post-extraction tissue healing in wisdom tooth Surgery: double-blind randomized clinical trial. Pain Manag. 2025 Sep;15(9):555-569. doi: 10.1080/17581869.2025.2528590. Epub 2025 Jul 5. PMID 40616597